CLINICAL TRIAL: NCT03396562
Title: The eXtroardinarY Babies Study: Natural History of Health and Neurodevelopment in Infants and Young Children With Sex Chromosome Trisomy
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0118
Record Dates: First submitted 2017-12-05; First posted 2018-01-11 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Klinefelter Syndrome; Trisomy X; XYY Syndrome; XXXY and XXXXY Syndrome; Xxyy Syndrome; Xyyy Syndrome; Xxxx Syndrome; Xxxxx Syndrome; Xxxyy Syndrome; Xxyyy Syndrome; Xyyyy Syndrome; Male With Sex Chromosome Mosaicism
Keywords: body composition; klinefelter syndrome; XXY; Trisomy X; XXX; XYY; XXYY; XXXY; XXXXY; sex chromosome variation; sex chromosome aneuploidy; sex chromosome trisomy; testosterone; XYYY; XXXX; XXXXX; XXXYY; XXYYY; XYYYY; developmental delay; speech development
MeSH Terms: conditions — Klinefelter Syndrome; Triple X syndrome; 47, XYY syndrome; Tetrasomy X; 49,XXXXX syndrome; Learning Disabilities | interventions — Growth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A venous blood, urine and stool samples will be collected at each research visit, with the exception of the 18 and 48 month visit.
  Hormone levels (Follicle Stimulating Hormone, Luteinizing Hormone, Anti-Mullerian Hormone, Inhibin B, Estradiol and Testosterone) will be analyzed. Some of the venous blood will be collected for the purpose of banking serum, plasma, RNA and DNA for future studies. Urine and stool samples will also be banked for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCT Conditions: Sex Chromosome Trisomies Conditions including Klinefelter (XXY), Trisomy X (XXX), XXY Syndromes.
  Interventions: Longitudinal observational assessments of development and growth at ages: 2 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, and 5 or 6 years.
  Interventions: Other: Assessments of Development and Growth

INTERVENTIONS:
Other: Assessments of Development and Growth — Longitudinal observational assessments of development and growth at ages: 2 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 5 years, 6 years, 7 years, 8 years, 9 years of age.

SUMMARY:
This study is designed to research the natural history of neurodevelopment, health and early hormonal function in infants with XXY/Klinefelter syndrome, XYY, XXX and other sex chromosome variations in an effort to identify early predictors of developmental and health outcomes. The Investigators will also evaluate different developmental screening tools in infants with sex chromosome variations so the investigators can develop recommendations for pediatrician caring for infants and young children with XXY/Klinefelter syndrome, XYY, XXX, and other sex chromosome variations.

DETAILED DESCRIPTION:
Background: Sex Chromosome Trisomies (SCT) including Klinefelter (XXY), Trisomy X (XXX), and XYY syndromes occur in 1 out of every 500 births and are associated with a broad phenotypic spectrum including increased risk for developmental delays (DD), language/learning disorders, and autism spectrum disorder (ASD). XXY is also associated with testicular failure, XXX increases risk for ovarian failure, and disorders of insulin resistance and other medical problems resulting in increased morbidity and mortality occur in all 3 SCTs. Historically, less than 10% of SCT diagnoses occur in childhood, however the rate of newborns with SCT has markedly increased with new noninvasive prenatal cell-free DNA (cfDNA) screening. SCT natural history research is limited to studies from the 1970's, and the investigators have little knowledge of early predictors of the wide heterogeneity in later outcomes. The high risk for DD in SCT suggests that newborn screening may improve identification for DD and timely initiation of interventions. However, it is not clear whether all SCT infants indeed require intensive developmental assessments and therapies, or if primary care screenings are sufficient to identify those in need. The surge in prenatal SCT diagnoses from cfDNA methods provides an opportunity for longitudinal study of a cohort of infants to explore natural history, and to improve care.

Aims: This study aims to: (1) describe and compare the natural history of neurodevelopment, health and early gonadal function in infants with the 3 SCT conditions through a national prospective eXtraordinarY Babies Study in partnership with the Newborn Screening Translational Research Network (NBSTRN), (2) identify early predictors of poor neurodevelopmental and cardiometabolic outcomes, and (3) evaluate the sensitivities of common primary care developmental screening measures to detect DD and ASD in this high-risk population to inform recommendations for an early neurodevelopmental care protocol.

Approach: Infants with a prenatal diagnosis of XXY, XYY, or XXX will be followed prospectively every 6-12 months for 2-4 years at 2 eXtraordinarY Kids Clinic sites. Demographics, health history, development, interventions, and social/family history will be collected. Assessments will include: (1) measures of cognitive, language, social, motor, and adaptive function, (2) physical exam, gonadal function labs, cardiometabolic measures, and body composition, and (3) quality of life outcomes. Impact: Prospective study of the natural history of prenatally diagnosed infants with SCT will allow investigation of important questions to inform newborn screening considerations, such as the interplay between early hormonal profiles and developmental outcomes. Results will be immediately relevant for counseling and establishing evidence-based care guidelines for the rapidly increasing rate of SCT diagnoses from cfDNA screening. Results will serve as the basis for ongoing longitudinal studies of health and psychological outcomes of SCTs through the lifespan.

ELIGIBILITY:
Inclusion Criteria:

1. Prenatal diagnosis of sex chromosome aneuploidy (by cfDNA, chorionic villi sampling, and/or amniocentesis)
2. Postnatal confirmatory karyotype of XXY, XYY, XXX, XXYY, XYYY, XXXY, XXXX, XXXXX, XXXXY, XXXYY, XXYYY, XYYYY (including any mosaicism with <80% 46,XX or 46,XY cell line)
3. English or Spanish speaking
4. Age 6 weeks to 12 months 30 days on enrollment

Exclusion Criteria:

1. Previous diagnosis of a different genetic or metabolic disorder with neurodevelopmental or endocrine involvement
2. Prematurity less than 34 weeks gestational age
3. Complex congenital malformation not previously associated with sex chromosome aneuploidy
4. History of significant neonatal complications (ie intraventricular hemorrhage, meningitis, hypoxic-ischemic encephalopathy)
5. Known complex Central Nervous System (CNS) malformation identified by neuroimaging

Ages: 6 Weeks to 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sex Chromosome Trisomies (SCT) including Klinefelter (XXY), Trisomy X (XXX), and XYY. Rare sex tetrasomy and pentasomy conditions are also eligible.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-09-29 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Descriptive Statistics of Cognitive Scores on the Bayley-III | 36 months
  Cognitive skills will be assessed using the standardized Bayley Scales of Infant Development--3rd Edition (Bayley-3)
Longitudinal Descriptive Statistics of Motor Scores on the Bayley-III | 36 months
  Motor development will be assessed using the standardized Bayley Scales of Infant Development--3rd Edition (Bayley-3)
Longitudinal Descriptive Statistics of Language Scores on Bayley-III | 36 months
  Language development will be assessed using the Bayley Scales of Infant Development--3rd Edition (Bayley-3)

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 36 months
  BMI will be determined through measurement of length and weight at the research visit.
Z Score | 36 months
  The z score will be calculated for age group at the research visit.
Body Composition (% body fat) | 3 year old visit
  Body fat percentage will be measured using air Dual Energy X-Ray Absorptiometry (DEXA) at 3 year old visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Tartaglia, MD MS, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours at Thomas Jefferson University, Philadelphia, Pennsylvania